CLINICAL TRIAL: NCT04709705
Title: Randomized Controlled Trial Comparing Dimethyl Sulfoxide Cryopreserved Platelets to Liquid Stored Platelets in Patients Undergoing Cardiopulmonary Bypass Surgery (CRYPTICS)
Brief Title: DMSO Cryopreserved Platelets in Cardiopulmonary Bypass Surgery (CRYPTICS)
Acronym: CRYPTICS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cellphire Therapeutics, Inc. (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-16-15
Record Dates: First submitted 2020-11-18; First posted 2021-01-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery
Keywords: Cryopreserved Platelets

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group, active comparator-controlled trial to evaluate the noninferiority or superiority of CPP with LSP in controlling blood loss in patients undergoing CPB surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryopreserved platelets (Experimental): Cryopreserved platelets to be given intraoperatively or post operatively up to 3 units post-heparin reversal
  Interventions: Biological: Human platelets
- Liquid stored platelets (Active Comparator): Liquid stored platelets to be given intraoperatively or post operatively up to 3 units post-heparin reversal
  Interventions: Biological: Human platelets

INTERVENTIONS:
Biological: Human platelets — Platelets given to control bleeding

SUMMARY:
A randomized, parallel group, active comparator-controlled trial to evaluate the non-inferiority or superiority of Cryopreserved Platelets with Liquid Stored Platelets in controlling blood loss in patients undergoing Cardiopulmonary Bypass Surgery.

DETAILED DESCRIPTION:
A randomized, parallel group, active comparator-controlled trial to evaluate the non-inferiority or superiority of Cryopreserved Platelets with Liquid Stored Platelets in controlling blood loss in patients undergoing Cardiopulmonary Bypass Surgery. Patients planning to undergo Cardiopulmonary Bypass Surgery with risk factors for significant bleeding post-surgery will be approached. Subjects will be randomized in a 1:1 ratio to receive either Cryopreserved Platelets or Liquid Stored Platelets. Eligible subjects will undergo Cardiopulmonary Bypass Surgery and at the completion of bypass and heparin reversal subjects will likely be assessed for eligibility before coming off bypass. Study platelets will be given either intraoperatively after heparin reversal and return of active clotting time (ACT) to < 140 sec or post operatively (after chest closure).

A single unblinded interim analysis on the primary efficacy endpoint will be performed for this study after 75% of the planned number of mITT subjects are treated (i.e., after 150 mITT subjects are treated, irrespective of the number of subjects in each treatment group).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age
2. Undergoing CPB surgery with at least one risk factor for post-surgical bleeding including:

   1. All re-operative cardiac procedures.
   2. Expected bypass > 120 minutes.
   3. Any combined cardiac surgery procedures (e.g. multiple valve, valve/CABG).
   4. Any procedure that in the estimation of the surgical attending, has a high likelihood of receiving platelets
3. Ability to comprehend and willingness to sign informed consent.
4. If female of childbearing potential, have a negative pregnancy test on the day of the surgery and prior to the surgery agrees to use a method of highly effective birth control from the time of consent through the end of the safety follow-up period (Day 6 or discharge from hospital, whichever is earlier). Note: women must have been surgically sterilized [bilateral tubal ligation, bilateral oophorectomy, total hysterectomy) or postmenopausal (≥50 years of age and continuous amenorrhea for 24 months) to be considered non-childbearing potential.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Undergoing any of the following surgical procedures:

   1. Coronary artery bypass surgery alone
   2. Implantation of ventricular assist device
   3. Thoracoabdominal aortic aneurysm repair
2. Known or suspected pregnancy or breastfeeding
3. History of any major unprovoked thrombotic events
4. History of heparin-inducted thrombocytopenia
5. Active infection treated with antibiotics
6. Refuse transfusion of blood products for religious or other reasons
7. Previous enrollment in this study
8. Immune thrombocytopenic purpura
9. Known allergy to DMSO
10. In the judgement of the investigator, is not a good candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint assessed from time zero until the drain tubes are removed or 24 hours post time zero. | From "time zero" until the drain tubes are removed or 24 hours post time zero, whichever is earlier
  Total volume of chest tube drainage assessed by measurement of the volume of blood collected from the mediastinal and pleural drains from "time zero", the time of 1) chest closure or equivalent, 2) chest tubes or equivalent are attached to a graduated post drainage system, and 3) with suction (defined as time zero for analytical purposes) determined in mL/kg every hour during the first 12 hours and at 6-hour intervals thereafter, for up to 24 hours or chest tube removal (whichever is earlier).

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint assessed from time zero until the drain tubes are removed or 24 hours post time zero. | From "time zero" until the drain tubes are removed or 24 hours post time zero, whichever is earlier
  The primary endpoint given in mL/kg
Secondary Efficacy Endpoint assessed at 6 hours interval through 24 hours post time zero or when the chest tubes are removed. | 6 hours intervals through 24 hours post time zero or when chest tubes are removed, whichever is earlier.
  Chest tube drainage volume (mL) collected at 6 hours intervals through 24 hours post time zero or tube removal, whichever is earlier.
Secondary Efficacy Endpoint at 6 hours intervals through 24 hours post time zero or when chest tubes are removed | 6 hours intervals through 24 hours post time zero or when chest tubes are removed, whichever is earlier
  Drainage rate (mL/hr) collected at 6 hours intervals through 24 hours post time zero or when chest tube are removed, whichever is earlier.
Secondary Efficacy Endpoint assessed at the end of first study platelet transfusion through 24-hour post heparin reversal (Efficacy follow-up period) | Infused after the end of the first study platelet transfusion through 24-hour post heparin reversal (Efficacy follow-up period)
  Total units by type of other post-operative blood products (pRBC, non-study platelets, CRYO, plasma, clotting factor concentrates) infused after the end of the first study platelet transfusion until end of the efficacy follow-up period
Secondary Efficacy Endpoint assessed within 24 hour post heparin reversal (Efficacy follow-up period) | Within the 24 hour period after heparin reversal
  Incidence of surgical re-exploration and incidence of verified surgical or other causes for bleeding within the 24 hour period after heparin reversal
Secondary Efficacy Endpoint assessed from first protamine administration to the time of first suture for incision closure on Day 1 (Day of Surgery) | Time from first protamine administration to the time when the surgeon initiates the first suture for incision closure, Day 1 (Day of operation)
  Time to hemostasis (defined as the time from first protamine administration to the time when the surgeon initiates the first suture for incision closure)
Secondary Efficacy Endpoint assessed at the first study platelet transfusion through 24-hour post heparin reversal (Efficacy follow-up period) | Time of first study platelet transfusion through 24-hour post heparin reversal (Efficacy follow-up period)
  Treatment failure (defined as requiring more than three units of study treatment (CPP or LSP))

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - University of Colorado, Aurora, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - UF Health, Gainesville, Florida
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State Univ. Wexner Medical Center, Columbus, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson Univ. Hospital, Philadelphia, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Cardiac Vascular, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No